CLINICAL TRIAL: NCT04491721
Title: Long-term Follow-up the OS and PFS of Rituximab Biosimilar HLX01 and MabThera in Combination With CHOP, in Previously Untreated Subjects With CD20+ DLBCL
Brief Title: Follow-up the OS and PFS of Rituximab Biosimilar HLX01 and MabThera, in Untreated Subjects With CD20+ DLBCL
Status: Enrolling by invitation | Type: Observational
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shi Yuankai, chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: NCC2288
Record Dates: First submitted 2020-07-25; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: rituximab; overall survival; progression-free survival
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Rituximab Biosimilar HLX01 in Combination With CHOP: Rituximab Biosimilar HLX01 in Combination With CHOP,in Previously Untreated Subjects With CD20+ DLBCL.
- MabThera in Combination With CHOP: MabThera in Combination With CHOP，in Previously Untreated Subjects With CD20+ DLBCL.

SUMMARY:
The main objective of this study is to observe the overall survival of Rituximab Biosimilar HLX01 and MabThera in Combination With CHOP, in previously untreated subjects with CD20+ DLBCL. The secondary objective of this study is to observe the progression-free survival of Rituximab Biosimilar HLX01 and MabThera in Combination With CHOP, in previously untreated subjects with CD20+ DLBCL.

DETAILED DESCRIPTION:
1. Enrollment:407 subjects.
2. The inclusion criteria of this study: subjects who have participated in Phase III clinical trials.Phase III clinical trial（NCT02787239） has ended.
3. The exclusion criteria: ①Subjects died; ②Subjects are unwilling to participate in follow-up study; ③ the investigator judges that the subject is not suitable for participating the study.
4. Duration and method of follow-up: 2-10 years (2020-2027)after the end of the Phase III trial and follow up the subjects by the phone.
5. Statistical analysis method: For progression-free survival and overall survival (OS), the median time and its 95% confidence intervals will be calculated by the Kaplan-Meier method.The Log-Rank test will be used for finding the difference between groups. The efficacy will be analyzed by SAS9.4 , and all hypothesis tests are two-sided. The confidence level of all confidence intervals is 95%. P value less than 0.05 was regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have participated in Phase III study（NCT02787239）.

Exclusion Criteria:

* ①Subjects died; ②Subjects are unwilling to participate in follow-up study; ③ the investigator judges that the subject is not suitable for participating the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have participated in Phase III study. Phase III study（NCT02787239）was rituximab biosimilar HLX01 and MabThera in patients with diffuse large B-cell lymphoma.
Sampling Method: Non-Probability Sample
Enrollment: 407 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
overall survival | up to 8 years
  The main objective of this study is to observe the overall survival of Rituximab Biosimilar HLX01 and MabThera in Combination With CHOP, in previously untreated subjects with CD20+ DLBCL.

SECONDARY OUTCOMES:
progression-free survival | up to 8 years
  The secondary objective of this study is to observe the progression-free survival of Rituximab Biosimilar HLX01 and MabThera in Combination With CHOP, in previously untreated subjects with CD20+ DLBCL.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Doctor, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, China